CLINICAL TRIAL: NCT06477965
Title: Multicenter National Registry for Artery Embolization (Embo Registry) for the Treatment of Osteoarthritis and Areas of Localized Pain to Assess Treatment of Artery Embolization to Determine If Subjects Have Decrease Pain, Decreased Use of Narcotics and NSAIDs, and Quality of Life Improvement Post Procedure.
Brief Title: Embo Registry; National Registry for Artery Embolization
Status: Recruiting | Type: Observational
Sponsor: Vascular Solutions of North Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 20241915
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain; Osteoarthritis, Knee; Osteoarthritis Thumb; Osteoarthritis Shoulder; Pain, Chronic; Tendonitis Elbow; Tendonitis Shoulder; Tendonitis;Achilles; Tenosynovitis
Keywords: Pain; Osteoarthritis; Arthritis; Tendonitis; Tenosynovitis
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee; Tenosynovitis; Pain; Osteoarthritis; Arthritis; Tendinopathy | interventions — Uterine Artery Embolization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group: For the study to determine efficacy and overall improvement of patients post artery embolization by comparing patient's pain preoperative and post operatively, if there is a decreased use of medication preoperatively compared to post procedure and increased quality of life preoperative and post procedure. Clinical outcomes of improvement will be determined by improvement of Visual Analog Scale (VAS) scores, Western Ontario and McMaster Universities Index (WOMAC), EQ-5D-5L Quality of Life Questionnaire, and to determine if patients had decrease used of medication prescribed preoperatively.
  Interventions: Procedure: Artery Embolization

INTERVENTIONS:
Procedure: Artery Embolization — Embolic Solution are intended for use in occluding blood vessels for therapeutic or operative purposes. The embolic solution is used during an outpatient procedure, the physician will insert a small catheter onto the artery supplying the lining of the target joint or target localized pain. Tiny particles are then injected through the catheter into these arteries, reducing blood flow to the target area. This reduces the amount of inflammation associated with osteoarthritis, tendonitis, tenosynovitis or an injury, a process that can help decrease symptoms or eliminate the associated localized pain to this area. With understanding that it does not treat the underlying cartilage destruction or underlying condition causing pain but would like to determine the efficacy and validity of this treatment.
  Other Names: Genicular Artery Embolization; GAE

SUMMARY:
Embo Registry is a retrospective and prospective observational study to evaluate real world effectiveness and the use of Artery Embolization as a treatment for chronic pain with patients that have osteoarthritis and localized pain to provide symptomatic relief. This study is to determine the efficacy and validity of procedure and that following procedure patients had decreased pain and improved quality of life.

DETAILED DESCRIPTION:
Embolic Solution are intended for use in occluding blood vessels for therapeutic or operative purposes. The embolic solution is used during an outpatient procedure, the physician will insert a small catheter onto the artery supplying the lining of the target joint or target localized pain. Tiny particles are then injected through the catheter into these arteries, reducing blood flow to the target area. This reduces the amount of inflammation associated with osteoarthritis, tendonitis, tenosynovitis or an injury, a process that can help decrease symptoms or eliminate the associated localized pain to this area. With understanding that it does not treat the underlying cartilage destruction or underlying condition causing pain but would like to determine the efficacy and validity of this treatment. For the study to determine efficacy and overall improvement of patients post procedure by comparing patient's pain preoperative and post operatively, if there is a decreased use of medication preoperatively compared to post procedure and increased quality of life preoperative and post procedure. Clinical outcomes of improvement will be determined by improvement of Visual Analog Scale (VAS) scores, Western Ontario and McMaster Universities Index (WOMAC), EQ-5D-5L Quality of Life Questionnaire, and to determine if patients had decrease used of medication prescribed preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age undergone artery embolization interventions for the treatment of chronic pain due to osteoarthritis or other diagnoses that cause localized pain.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic and localized pain from diagnoses such as osteoarthritis, tendonitis, tenosynovitis, or injury who underwent Artery Embolization for the treatment of their symptoms/pain.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 3 months
  Clinical success at 3 months, defined as improvement in Western Ontario and McMaster University (WOMAC) Pain Subscale from pre-operative/baseline WOMAC scores.
Primary Outcome | 3 months
  Clinical success at 3 months, defined as improvement of Visual Analog Scale (VAS) Scores from pre-operative/baseline scores.
Primary Outcome | 3 months
  Comparative assessment at 3 months of decreased use of medication prescribed at baseline to 3 months post operatively.
Primary Outcome | 3 months
  Clinical success at 3 months, as defined by improvement in the quality of life using the EQ-5D-5L Quality of Life Questionnaire compared to baseline.

SECONDARY OUTCOMES:
Secondary Outcome | 12 months
  Number of patients achieving clinical success at 1,3, 6, and 12-months post procedure.
Secondary Outcome | 12 months
  Decrease in Western Ontario and McMaster University (WOMAC) index compared to baseline, 1, 3, 6, and 12 months.
Secondary Outcome | 12 months
  Pain score assessed using Visual Analog Scale (VAS) Score from baseline, 1, 3, 6, and 12 months.
Secondary Outcome | 12 months
  Number of subjects who had pain reduction >50% in the mean VAS pain scale at 1, 3, 6 and 12 months in comparison with baseline/preprocedural assessments.
Secondary Outcome | 12 months
  Change in the use of narcotics or non-steroidal anti-inflammatory drugs (NSAID's) compared to baseline through 1, 3, 6, and 12 months.
Secondary Outcome | 12 months
  Change in quality of life using the EQ-5D-5L Quality of Life Questionnaire compared to baseline through 1, 3, 6, and 12 months.
Secondary Outcome | 12 months
  Number of patients with confirmed cases of osteoarthritis with a Kellgren and Lawerence Grade Level 2-3 (confirmed by X-Ray) improved symptoms compared to baseline through to 1, 3, 6 and 12-months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Rao, MD, Principal Investigator — Vascular Solutions of North Carolina; Amer Iqbal, Study Director — Vascular Solutions of North Carolina; Meaghan Thomas, CCRP, Study Chair — Vascular Solutions of North Carolina
Locations (2):
- United States (2):
  - Vascular Solutions of North Carolina, Cary, North Carolina
  - Southern Tennessee Cardiology, Winchester, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Dissemination of data will be through publications in peer-reviewed scientific journals, national and international meeting, on-line presentations, and providing de-identified data to participating site investigators and by providing analysis results upon request from site investigators.
Supporting Information: CSR
Time Frame: 12 months
Access Criteria: Must contact sponsor for approval or participate in study research.
URL: https://emboregistry.ai

REFERENCES:
- See also: contact study — https://emboregistry.ai